CLINICAL TRIAL: NCT01629160
Title: Characterization of Normal and Abnormal Ventricular Wall Motion
Brief Title: Ventricular Wall Motion Characterization
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: 642
Record Dates: First submitted 2012-06-24; First posted 2012-06-27 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Atrial Fibrillation; Tachycardia, Ventricular
MeSH Terms: conditions — Atrial Fibrillation; Tachycardia, Ventricular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to evaluate feasibility of using new technologies to characterize ventricular wall motion in patients indicated for mapping and ablation procedures. Echo will be performed preoperatively and patients will receive a 1-month followup telephone call.

ELIGIBILITY:
Inclusion Criteria:

* Be in sinus rhythm
* Have the ability to provide informed consent for study participation and be willing and able to comply with the Clinical Investigational Plan described evaluations
* Be undergoing mapping and ablation that requires left heart access for either ventricular tachycardia (VT) or atrial fibrillation (AF) according to HRS (Heart Rhythm Society)/ESC (European Society of Cardiology)/German National guidelines. The patient needs to have at least one of the following indications for left heart mapping and ablation to be included in the study: a) Symptomatic sustained monomorphic VT (SMVT), or b) Frequent PVCs, non-sustained VT, or VT that is presumed to cause ventricular dysfunction, or c) Bundle branch reentrant or interfascicular VTs, or d) Symptomatic AF with indication for ablation per current HRS/ESC/German National guidelines in a patient who is either 1) refractory or intolerant to at least one Class 1 or Class 3 antiarrhythmic medication, or 2) unable/unwilling to take antiarrhythmic drug therapy and chooses ablation as the first line of therapy

Exclusion Criteria:

* Have permanent AF
* Exhibit Cheyne-Stokes respiration
* Have a recent myocardial infarction within 40 days prior to enrollment
* Have undergone cardiac surgery or coronary revascularization procedure within 3 months prior to enrollment or be scheduled for such procedures
* Have had a recent CVA or TIA within 3 months prior to enrollment
* Be less than 18 years of age
* Be pregnant
* Be currently participating in any other clinical investigation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Atrial Fibrillation or Ventricular Tachycardia
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2012-07; Primary Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Feasibility of Ventricular Wall Motion Characterization | Mapping and Ablation Procedure

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Hindricks, MD, Principal Investigator — Herzzentrum Leipzig GmbH
Locations (1):
- Herzzentrum Leipzig GmbH, Leipzig, Germany

REFERENCES:
- [Derived] Piorkowski C, Arya A, Markovitz CD, Razavi H, Jiang C, Rosenberg S, Breithardt OA, Rolf S, John S, Kosiuk J, Huo Y, Doring M, Richter S, Ryu K, Gaspar T, Prinzen FW, Hindricks G, Sommer P. Characterizing left ventricular mechanical and electrical activation in patients with normal and impaired systolic function using a non-fluoroscopic cardiovascular navigation system. J Interv Card Electrophysiol. 2018 Apr;51(3):205-214. doi: 10.1007/s10840-018-0317-3. Epub 2018 Jan 31. PMID 29388068